CLINICAL TRIAL: NCT01331954
Title: Treatment of Breast Fibroadenoma With High Intensity Focused Ultrasound (HIFU): a Feasibility Study
Brief Title: Treatment of Breast Fibroadenoma With High Intensity Focused Ultrasound (HIFU)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU/BG/FA/Jan2011
Record Dates: First submitted 2011-04-07; First posted 2011-04-08 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Breast Fibroadenoma
MeSH Terms: conditions — Fibroadenoma

ARMS (1):
- HIFU (Experimental)
  Interventions: Device: Ultrasonic ablation device

INTERVENTIONS:
Device: Ultrasonic ablation device — One or two HIFU procedures
  Other Names: TH-One

SUMMARY:
Demonstrate the efficacy of High Intensity Focused Ultrasound in the treatment of the breast fibroadenoma.

ELIGIBILITY:
Inclusion Criteria:

* One breast fibroadenoma with diagnosis based on:

  * Clinical examination
  * Ultrasound image
  * For women older than 35 years: mammogram with BI-RADS score < 3
  * Histologic confirmation by two independent readers
* Fibroadenoma size between 1 cm and 3 cm at its largest dimension (measured by ultrasound)

Exclusion Criteria:

* Patient pregnant or lactating
* Bi-RADS score > 2 at the mammogram, or microcalcifications within the lesion.
* History of breast cancer or history of laser or radiation therapy to the target breast
* Breast implants
* Breast cyst
* Fibroadenoma not clearly visible on the ultrasound images (in B mode)
* Patient participating in other trials using drugs or devices

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-03 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Reduction of breast fibroadenoma volume at ultrasonography | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roussanka Kovatcheva, M, Principal Investigator — University Hospital of Endocrinology (USBALE) "Acad. Ivan Penchev"
Locations (1):
- University Hospital of Endocrinology (USBALE) "Acad. Ivan Penchev", Sofia, Bulgaria

REFERENCES:
- [Derived] Kovatcheva R, Zaletel K, Vlahov J, Stoinov J. Long-term efficacy of ultrasound-guided high-intensity focused ultrasound treatment of breast fibroadenoma. J Ther Ultrasound. 2017 Mar 16;5:1. doi: 10.1186/s40349-017-0083-1. eCollection 2017. PMID 28331611